CLINICAL TRIAL: NCT06264388
Title: A Biomarker-Guided Phase 2 Study of DB107-RRV (Retroviral Replicating Vector) Combined With DB107-Flucytosine Extended-Release Tablets in Patients With Recurrent Glioblastoma or Anaplastic Astrocytoma
Brief Title: DB107-Retroviral Replicating Vector (RRV) Combined With DB107-Flucytosine (FC) in Patients With Recurrent Glioblastoma or Anaplastic Astrocytoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ashish Shah (Other)
Collaborators: Denovo Biopharma LLC (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Ashish Shah, Assistant Professor of Clinical, University of Miami
Organization: University of Miami (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20231234; R21CA282543 (NIH)
Record Dates: First submitted 2024-02-08; First posted 2024-02-20 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: High Grade Glioma; Anaplastic Astrocytoma
MeSH Terms: conditions — Glioma; Astrocytoma | interventions — Flucytosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- DB107-RRV and DB107-FC Group (Experimental): Patients will receive DB107-RRV during the tumor resection/biopsy procedure. Approximately 6 weeks after surgery, patients will start drug therapy with a 7-day oral regimen of 220 mg/kg/day DB107-FC, which is to be self-administered. This 7-day regimen, which is considered one cycle of treatment, is to be repeated every 6 weeks for up to 12 months. Patients will undergo follow up procedures for at least 5 years after last DB107-RRV treatment.
  Interventions: Drug: DB107-RRV; Drug: DB107-FC

INTERVENTIONS:
Drug: DB107-RRV — Patients will undergo surgery to remove as much of the high-grade glioma (HHG) tumor as possible and will receive combination intravenous (IV) and adaptive repeat intratumoral delivery of DB107-RRV in the vein (IV) and in the walls of the cavity that remains where tumor is removed.
Drug: DB107-FC — Patients will start taking DB107-FC three times by mouth every day for a period of seven days, which is one cycle of treatment. A cycle of treatment is medication taken on a set schedule with periods of rest in between. Patients will wait five weeks before taking the next seven day course of DB107-FC. The first dose of DB107-FC will be taken at the hospital or clinic; afterward, patients will take the doses of DB107-FC at home. Patients will take DB107-FC for up to 12 months after surgery.
  Other Names: Ancobon; Ancotil

SUMMARY:
The purpose of this study is to determine if the investigational products, DB107-RRV and DB107-FC, as a combination treatment will shrink high-grade glioma (HGG) in patients with recurrent/progressive, resectable or unresectable disease and increase the time that disease is controlled.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18-75 years old.
2. Histologically proven HGG that have recurred/progressed (first or second recurrence).
3. Patients with unresectable or resectable HGG (AA or GBM) will be enrolled.
4. Measurable disease on MRI as evidenced by 1 cm on two separate dimensions on MRI fluid attenuated inversion recovery (FLAIR) (non-enhancing) or contrast-enhancement.
5. Last temozolomide dosage 4 weeks prior to surgery.
6. Patients with prior radiation therapy are allowed, but histological tumor diagnosis of recurrent tumor must be confirmed according to the RANO criteria. Recurrence must be confirmed by diagnostic biopsy with local pathology review or contrast-enhanced MRI. If first recurrence of GBM is documented by MRI, an interval of at least 12 weeks after the end of prior radiation therapy is required unless there is either: i) histopathologic confirmation of recurrent tumor, or ii) new enhancement on MRI outside of the radiotherapy treatment field.
7. Presence of Denovo Genomic Marker 7 (DGM7) biomarker in blood.
8. Laboratory values (Platelet count ≥ 80,000, hemoglobin [Hg] ≥10 g/dL, absolute neutrophil count (ANC) > 1,500 cells/mm3, absolute lymphocyte count (ALC) > 500/mm3) and adequate liver function, total bilirubin< 1.5 upper limit of normal (ULN), alanine transaminase (ALT) <2.5 ULN. Estimated glomerular filtration rate (eGFR) should be > 50 mL/min (Cockcroft Gault Formula). Patients with aspartate transaminase (AST) or ALT values >3 ULN and total bilirubin >1.5 mg/dL will be excluded.
9. Patients cannot be pregnant at the time of enrollment or during the study. Patients willing to use one (1) effective method of contraception in addition to barrier methods (condoms) from the time of signing the informed consent form until 12 months after receiving the last dose of DB107-RRV or until there is no evidence of DB107-RRV in their blood, whichever is longer.
10. Karnofsky Performance Score (KPS) ≥ 70.
11. Patient is able to consent and abide by protocol.

Exclusion Criteria:

1. History of active other malignancy (other than non-melanoma skin cancers, cervical ductal carcinoma in situ or localized prostate cancer) within 5 years.
2. Multifocal gliomas that cannot undergo stereotactic biopsy/administration of DB107-RRV will be excluded. Patients with 3 or more intracranial recurrences will be excluded.
3. Histologically confirmed oligodendroglioma or mixed gliomas.
4. History of human immunodeficiency virus (HIV) infection or other forms of severe immunosuppression.
5. Patients with impaired renal function (eGFR<50 cc/min).
6. Patients with bone marrow depression, such as those with a hematological disease or who are being treated with radiation or drugs that depress bone marrow or individuals who have a history of treatment with drugs or radiation that depress bone marrow within 1 month of enrollment.
7. The patient intends to undergo treatment with the Gliadel® wafer at the time of this surgery or has received the Gliadel® wafer < 30 days from surgery.
8. Allergy to 5-FC.
9. Gastrointestinal diseases that prevent absorption of medications such as 5-FC.
10. Pregnancy or patients who are actively breast-feeding.
11. Recent use of cytosine arabinoside (< 3 weeks).
12. Recent treatment with bevacizumamab (< 3 weeks).
13. Recent treatment with temozolomide (<4 weeks).
14. History of bleeding diathesis or current anti-coagulant or anti-platelet usage, including nonsteroidal anti-inflammatory drugs (NSAIDs), at the time of the scheduled resection that cannot be stopped for surgery.
15. Sustained dependence on systemic dexamethasone (>8 mg/day) one month prior to surgery.
16. Severe systemic illnesses including cardiopulmonary dysfunction (New York Heart Association > Grade 2 congestive heart failure (CHF), uncontrolled arrhythmias, significant pulmonary disease > Grade 2 dyspnea) or other serious medical condition or social situations that in the judgement of the Investigator(s) would interfere or limit compliance with study requirements/treatments.
17. The patient has or had any active infection requiring systemic antibiotic, antifungal or antiviral therapy within the past 4 weeks.
18. Current or active coronavirus disease (COVID-19) disease, positive quantitative polymerase chain reaction (qPCR) result.
19. Patients with impaired decision-making capacity.
20. Patients who are currently receiving investigational medications or medical device(s) within 4 weeks (or 5 half-lives of the investigational medication(s), whichever is shorter) prior to enrollment.
21. Patients who have any other disease, either metabolic or psychological, which as per Investigator assessment may affect the patient's compliance or place the patient at higher risk of potential treatment complications.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2034-05-01 (Estimated); Study Completion 2034-05-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | Up to 24 Months
  Progression free survival (PFS) is defined as duration from initiation of treatment to the point of disease progression or death.
Overall Survival | Up to 24 Months
  Overall survival (OS) refers to the duration from the initiation of enrollment until death, regardless of the cause.

SECONDARY OUTCOMES:
Assessment of Tumor Status Measured by Response Assessment in Neuro-oncology (RANO) Criteria | Up to 5 Years
  To evaluate the radiological response in participants with recurrent HGG based on overall response (CR) or partial response (PR), stable disease (SD), and progressive disease (PD) per the Response Assessment in Neuro-oncology (RANO) criteria.
Number of Treatment Related Toxicities | Up to 5 Years
  Number of treatment related toxicities will be assessed by the development of treatment-related ≥ Grade 3 adverse events as defined by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0.
Durable Response Rate (DRR) | Up to 5 Years
  Durable response rate (DRR) is defined as the proportion of patients whose best response to treatment is either complete response (CR) or partial response (PR) lasting at least 24 weeks as evidenced by MRI. DDR is calculated as the total number of patients with CR or PR lasting at least 24 weeks.
Durable Clinical Benefit Rate (DCBR) | Up to 5 Years
  Durable clinical benefit rate (DCBR) is defined as the proportion of patients whose best overall response is either CR or PR lasting at least 24 weeks or SD lasting at least 12 months according to modified RANO criteria as evidenced by MRI imaging. Durable clinical benefit rate is calculated as the total number of patients with CR or PR ≥ 24 weeks or with SD > 12 months.
Duration of Durable Response Rate | 12 Months
  Duration of durable response (DDR) is the tabulation of the total number of patients with CR, PR, SD, and PD at 12 months after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Ashish Shah, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami Hospital, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No